CLINICAL TRIAL: NCT00227526
Title: Enhancing Outcomes After Colon Surgery: Role of Prehabilitation Facilitating the Recovery Process.
Brief Title: Enhancing Outcomes After Colon Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Anesthesiologists' Society (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC02-053
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Surgery
Keywords: Colon; Surgery; Prehabilitation; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Prehabilitation

SUMMARY:
Most patients find that recovering from surgery is difficult particularly after abdominal surgery for cancer or other intestinal disorders. The surgical stress, healing process and concerns if further treatments are required suggest that the post-operative period may not be the best time to get people to exercise to rehabilitate lost functions. Prehabilitation is the process of enhancing functional capacity of the individual to enable him or her to withstand an incoming stressor, such as surgery, and this study aims to evaluate the effectiveness of prehabilitation for colorectal surgery. Two groups will be formed by a random process and the prehabilitation group will use an exercise cycle and weights to build endurance and strength for a 3-week period prior to surgery. The other group will receive training about exercises that will help them move better after surgery. People who are malnourished prior to surgery will receive nutritional supplements. The results of this trial will be used to inform practitioners and patients alike of the benefits (or risks if any) of exercise in preparing for surgery.

DETAILED DESCRIPTION:
The surgical process is a major stressor because of the psychological distress, tissue trauma, lack of activity, and quasi-starvation and it produces immediate systemic changes and both short- and long-term effects on activity and quality of life. However, there is mounting evidence that many of the negative immediate effects of surgery such as pain, fatigue, and weakness are amenable to intervention. If proper interventions are carried out, these symptoms may be readily controlled allowing for a faster recovery and early home discharge. But the effects of surgery are felt far beyond the immediate convalescent period and patients can feel fatigued for many weeks and this delays return to usual function and reduces quality of life. Thus, it would be of great practical benefit if ways of improving post-surgery physical function and quality of life could be identified.

Traditionally efforts have been made to improve the recovery process by intervening in the post-operative period. However, the post-operative period may not be the most opportune time to introduce interventions to accelerate recovery. Many of these surgical patients are concerned about perturbing the healing process as well as being depressed and anxious if they await further treatment. The pre-operative period may be a more emotionally salient time to intervene in the factors that contribute to recovery. The process of enhancing functional capacity of the individual to enable him or her to withstand an incoming stressor has been termed prehabilitation The purpose of this study is to address the following research question: Among persons scheduled for colorectal surgery, does a pre-operative program of aerobic and muscle strength training (prehabilitation) compared to a standard peri-operative educational protocol affect functional exercise capacity and health-related quality of life? The trial will be a single blind, stratified (on cancer diagnosis or not), randomized, two-group (prehabilitation or standard care), parallel design. Both groups will receive the same peri-operative education program. In conformity with current practice, all subjects will also be advised on nutritional support during the preoperative period. Persons with albumin < 38 gm./l will receive an adequate supply of protein and calorie nutritional supplement bars. In addition to this standard care, the prehabilitation group will be prescribed a program of exercise training consisting of daily stationary cycling from the start of the intervention to the day prior to surgery (minimum 3 weeks) combined with an individualized program of muscle strength training.

Both groups will be evaluated for exercise tolerance, walking capacity and health and emotional status at enrolment and after 3 three weeks of training as well as at 4 weeks, 8 weeks and 24 weeks (6 months) post-surgery. The main outcome measure will be the 6 Minute Walk Test - a valid and reliable measure of functional walking capacity. The estimator of effect will be the proportion of people in each group who, at 8 weeks post-surgery, achieve or exceed their baseline value on this test (± 20m). The proposed sample size is 200. This is based on 80% power to detect a difference of 22% in the proportion recovering to baseline values (40% in standard and 62% in prehabilitation). The results of this trial will be used to inform practitioners and patients alike of the benefits (or risks if any) of exercise in preparing for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Referred electively for colorectal resection for benign (polyposis adenoma diverticulitis) or non-disseminated colon and rectum cancers
* Referred electively for colorectal resection for colon reconstruction for non-active inflammatory bowel disease
* Referred electively for colorectal resection for fibrostenotic conditions that are a feature of Crohn's disease.

Exclusion Criteria:

* People with American Society of Anesthesiologists health status class 4-5
* Co-morbid medical conditions interfering with the ability to participate in either group or complete the testing procedures (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis)
* Patients at high risk for a cardiac complication during exercise at home: severe aortic stenosis, cardiac failure Class IV NYHA, myocardial infarction within 6 months, congestive heart failure, and unstable angina
* Persons with sepsis; and treatment with chemotherapy or radiotherapy during six months prior to the date of surgery
* Those with very low exercise tolerance (<3.5 METS) as determined by the baseline exercise test
* Anyone with a cardiac arrhythmia that manifests during the baseline exercise testing, prior to randomization
* Those people who are already in excellent physical condition owing to a regular participation in a high intensity physical activity. On testing, persons whose age-predicted value on the 6MWT exceeds 130% will be excluded (expected <10%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks

SECONDARY OUTCOMES:
V02 max and submax | baseline, 24 weeks
SF-36 - Short form 36 | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
CHAMPS - Community Healthy Activities Model Program for Seniors | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
Hospital Anxiety Depression Scale - HADS | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
Fatigue and Pain VAS | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
Visual Analogue Mood States (VAMS) | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
2Minute Walk Test | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
Complications: infection (wound, sepsis, urinary, lung); bleeding; wound dehiscence; technical complications (ileus, anastomotic leakage); stroke, MI, DVT/PE, delirium, fall w/wo injury; malnutrition; urinary retention; respiratory failure | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks
Charges for bed day: surgical procedure; surgeon/anaesthesiologist; pre, post and follow-up tests and procedures; visits; follow-up medications | baseline, 3 weeks, 4 weeks, 8 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Nancy Mayo, PhD, Principal Investigator — McGill University
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Carli F, Mayo N. Measuring the outcome of surgical procedures: what are the challenges? Br J Anaesth. 2001 Oct;87(4):531-3. doi: 10.1093/bja/87.4.531. No abstract available. PMID 11878719
- [Background] Carli F. Perioperative factors influencing surgical morbidity: what the anesthesiologist needs to know. Can J Anaesth. 1999 May;46(5 Pt 2):R70-9. doi: 10.1007/BF03013183. No abstract available. English, French. PMID 10370832
- [Background] Carli F, Mayo N, Klubien K, Schricker T, Trudel J, Belliveau P. Epidural analgesia enhances functional exercise capacity and health-related quality of life after colonic surgery: results of a randomized trial. Anesthesiology. 2002 Sep;97(3):540-9. doi: 10.1097/00000542-200209000-00005. PMID 12218518
- [Derived] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Derived] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503